CLINICAL TRIAL: NCT04201886
Title: Serum Calprotectin Level in Patients With Rheumatoid Arthritis and Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Badr, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: calprotectin in RA and OA
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis and Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RA patients (Other): A. Full history taking B. Physical examination C. Laboratory investigation: • Serum Calprotectin (CLP)
  Interventions: Other: serum calprotectin
- OA patients (Other): A. Full history taking B. Physical examination C. Laboratory investigation: • Serum Calprotectin (CLP)
  Interventions: Other: serum calprotectin

INTERVENTIONS:
Other: serum calprotectin — serum calcium binding leucocyte protein

SUMMARY:
Assessment of the serum level of calprotectin in patients with rheumatoid arthritis and osteoarthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory autoimmune disease with genetic susceptibility. It is characterized by chronic synovitis and progressive joint destruction. There is synovial infiltration by inflammatory cells, activation of synovial fibroblasts, and production of a wide range of inflammatory cytokines. Sustained high disease activity results in a poor disease outcome so assessment of inflammatory activity in RA is of pivotal importance for the optimal treatment in these patients. Disease activity of RA patients is assessed by clinical examination, laboratory tests and radiographic assessment (e.g. ultrasonography). Laboratory assessment of RA activity is done routinely by measuring acute phase reactants such as an erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP), which are elevated in most patients with RA. It has been demonstrated that more than 40% of RA patients have normal ESR or CRP (false negative results). Therefore, new serum markers that can more accurately reflect real inflammatory activity in RA patients are needed. Calprotectin (CLP) is a calcium binding leucocyte protein consisting of the heterocomplex of S100A8/ A9 (myeloid-related protein, MRP8/MRP14), as well as being a major monocyte/macrophage protein which has gained interest as a marker of inflammation in RA. Calprotectin has been identified as an important endogenous alarmin, one of the damage-associated molecular pattern (DAMP) molecules that acts as a ligand for the TLR4 receptor and amplifies the inflammation cascade via NF-kB and p38 mitogen-activated protein kinase. Calprotectin levels are higher in the serum of RA patients compared with healthy subjects or patients with osteoarthritis (OA), Still, no cut-off levels have been identified to help in the diagnosis of RA. Calprotectin is involved in cartilage damage in OA. Synovial lining macrophages play a role in the OA process and in cartilage damage. Moderate calprotectin increase has been observed in the serum of OA patients compared with healthy controls also serum calprotectin levels were found higher in OA patients with synovial inflammation compared with those without.

ELIGIBILITY:
Inclusion Criteria:

1. Adult RA Patients who fulfilled the 2010 ACR/European league against rheumatism (EULAR) criteria for the classification of RA
2. Adult osteoarthritis patients who fulfilled 2016 ACR revised Criteria for early diagnosis of knee OA

Exclusion Criteria:

1. Individuals with other autoimmune diseases (systemic lupus erythematosus, polyarteritis nodosa, dermatomyositis, scleroderma, spondyloarthritis, behcet's disease, psoriasis and inflammatory bowel disease).
2. RA patients with interstitial lung disease (IPF).
3. Patients with malignancy.
4. Patients with end stage organ failure.
5. Other conditions that may affect the serum level of calprotectin as diabetes mellitus, coronary artery disease, hepatitis and concomitant inflammatory disease as acute infection or chronic inflammatory status.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
• Assessment of sensitivity and specificity of the serum calprotectin as an indicator of disease activity in both RA and OA patients. | a year
  Analysis of serum level of calprotectin in both Rheumatoid arthritis and Osteoarthritis patients as an indicator of disease activity

SECONDARY OUTCOMES:
Compare between sensitivity and specificity of the serum calprotectin in detecting the activity of disease in both RA (Autoimmune inflammatory disease) and OA (Degenerative inflammatory disease) | a year
  Compare between sensitivity and specificity of the serum calprotectin in detecting the activity of disease in both RA (Autoimmune inflammatory disease) and OA (Degenerative inflammatory disease)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Hussien Abd El-Samea, Dr., Principal Investigator — Assiut university hospitals

REFERENCES:
- [Background] •Salehi Abari and Iraj. 2016 ACR revised criteria for early diagnosis of knee osteoarthritis. Autoimmune diseases and therapeutic approaches 2016; 3. 118.
- [Result] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Result] Copsey B, Thompson JY, Vadher K, Ali U, Dutton SJ, Fitzpatrick R, Lamb SE, Cook JA. Problems persist in reporting of methods and results for the WOMAC measure in hip and knee osteoarthritis trials. Qual Life Res. 2019 Feb;28(2):335-343. doi: 10.1007/s11136-018-1978-1. Epub 2018 Sep 18. PMID 30229533
- [Result] Hurnakova J, Hulejova H, Zavada J, Hanova P, Komarc M, Mann H, Klein M, Sleglova O, Olejarova M, Forejtova S, Ruzickova O, Vencovsky J, Pavelka K, Senolt L. Relationship between serum calprotectin (S100A8/9) and clinical, laboratory and ultrasound parameters of disease activity in rheumatoid arthritis: A large cohort study. PLoS One. 2017 Aug 23;12(8):e0183420. doi: 10.1371/journal.pone.0183420. eCollection 2017. PMID 28832684
- [Result] Hurnakova J, Hulejova H, Zavada J, Komarc M, Hanova P, Klein M, Mann H, Sleglova O, Olejarova M, Forejtova S, Ruzickova O, Vencovsky J, Pavelka K, Senolt L. Serum Calprotectin Discriminates Subclinical Disease Activity from Ultrasound-Defined Remission in Patients with Rheumatoid Arthritis in Clinical Remission. PLoS One. 2016 Nov 10;11(11):e0165498. doi: 10.1371/journal.pone.0165498. eCollection 2016. PMID 27832086
- [Result] Hurnakova J, Hulejova H, Zavada J, Komarc M, Cerezo LA, Mann H, Vencovsky J, Pavelka K, Senolt L. Serum calprotectin may reflect inflammatory activity in patients with active rheumatoid arthritis despite normal to low C-reactive protein. Clin Rheumatol. 2018 Aug;37(8):2055-2062. doi: 10.1007/s10067-018-4091-5. Epub 2018 Apr 14. PMID 29656372
- [Result] Douglas-Withers J, McCulloch K, Waters D, Parker K, Hogg N, Mitsuhashi T, Treharne GJ, Abbott JH, Stebbings S. Associations between Health Assessment Questionnaire Disability Index and physical performance in rheumatoid arthritis and osteoarthritis. Int J Rheum Dis. 2019 Mar;22(3):417-424. doi: 10.1111/1756-185X.13460. Epub 2018 Dec 17. PMID 30560589
- [Result] Jonsson MK, Sundlisaeter NP, Nordal HH, Hammer HB, Aga AB, Olsen IC, Brokstad KA, van der Heijde D, Kvien TK, Fevang BS, Lillegraven S, Haavardsholm EA. Calprotectin as a marker of inflammation in patients with early rheumatoid arthritis. Ann Rheum Dis. 2017 Dec;76(12):2031-2037. doi: 10.1136/annrheumdis-2017-211695. Epub 2017 Aug 16. PMID 28814431
- [Result] Kumar BS, Suneetha P, Mohan A, Kumar DP, Sarma KVS. Comparison of Disease Activity Score in 28 joints with ESR (DAS28), Clinical Disease Activity Index (CDAI), Health Assessment Questionnaire Disability Index (HAQ-DI) & Routine Assessment of Patient Index Data with 3 measures (RAPID3) for assessing disease activity in patients with rheumatoid arthritis at initial presentation. Indian J Med Res. 2017 Nov;146(Supplement):S57-S62. doi: 10.4103/ijmr.IJMR_701_15. PMID 29578196
- [Result] Mansour HE, Abdullrhman MA, Mobasher SA, El Mallah R, Abaza N, Hamed F, Khalil AAF. Serum Calprotectin in Rheumatoid Arthritis: A Promising Diagnostic Marker, How Far Is It Related to Activity and Sonographic Findings? J Med Ultrasound. 2017 Jan-Mar;25(1):40-46. doi: 10.1016/j.jmu.2016.11.001. Epub 2017 Jan 3. PMID 30065453
- [Result] Ometto F, Friso L, Astorri D, Botsios C, Raffeiner B, Punzi L, Doria A. Calprotectin in rheumatic diseases. Exp Biol Med (Maywood). 2017 Apr;242(8):859-873. doi: 10.1177/1535370216681551. Epub 2016 Jan 1. PMID 27895095
- [Result] Pincus T, Summey JA, Soraci SA Jr, Wallston KA, Hummon NP. Assessment of patient satisfaction in activities of daily living using a modified Stanford Health Assessment Questionnaire. Arthritis Rheum. 1983 Nov;26(11):1346-53. doi: 10.1002/art.1780261107. PMID 6639693
- [Result] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570